CLINICAL TRIAL: NCT05024149
Title: Assessing the Impact of Electroacupuncture on Facial Thermal Characteristics of Major Depressive Disorder Patients Based on Infrared Thermal Imaging Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Li, Attending Doctor, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020YKJ04
Record Dates: First submitted 2021-08-12; First posted 2021-08-27 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Major Depressive Disorder; Infrared Thermography
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy group (Experimental): Subjects in this group will not undergo acupuncture intervention. For participants in the healthy control group, the IRT examination of the measurement sites will last for 3 minutes, with one thermal image taken every 10s. In the Healthy group, there will be two visits, and the first visit will be considered as the screening stage (i.e., demographic data recording, medical history taking, physical examination report review and recording on the day of enrollment) and the second visit will be considered as the detection stage (i.e., the day of enrollment). At the second visit, the subjects received the Self-rating depression scale (SDS), HAMD, and then the infrared thermographic images to be acquired.
  Interventions: Other: infrared thermography (IRT)
- MDD electroacupuncture intervention group (Experimental)
  Interventions: Other: infrared thermography (IRT)
- MDD waiting-list group (Experimental): In this study, we used a waiting list control group. During the 4 weeks follow-up period, participants from the MDD waiting-list group had no contact with participants from the MDD EA intervention group and no access to the EA intervention. After the 4 weeks follow-up period, patients in the waiting list group received access to the EA intervention.
  Interventions: Other: infrared thermography (IRT)

INTERVENTIONS:
Other: infrared thermography (IRT) — The temperature and infrared thermography (IRT) images of the facial acupoints of three groups will be recorded by an infrared thermal-imaging camera.

SUMMARY:
Three groups of subjects will be included: 20 subjects in the healthy control group, 20 subjects in the MDD electroacupuncture (EA) intervention group, and 20 subjects in the MDD waiting-list group (participants will receive no treatment within 4 weeks). The temperature and infrared thermography (IRT) images of the facial acupoints of three groups will be recorded by an infrared thermal-imaging camera. The average facial temperature and acupoints temperature will be analyzed and compared within 3 groups. In addition, the correlation between facial infrared radiation characteristics of MDD patients and emotional changes will be explored. Besides, the relative specificity of the two meridians will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects:

1. Healthy subjects should provide a physical examination report within the last year, which could confirm they had not major systemic diseases, such as cardiovascular, respiratory, digestive, urinary, hematological, endocrine and neurological disease;
2. 18 ≤ age ≤ 60 years, both gender;
3. Subjects have clear consciousness and could communicate with others normally;
4. Subjects could understand the full study protocol and written informed consent is provided by themselves. Note: Subjects who meet the above four items will be included.

Inclusion criteria for MDD patients:

1. Meeting the above diagnostic criteria for MDD;
2. PHQ-9 score of 5 to 14, HAMD score of 21 to 35, and a diagnosis of mild or moderate depression by a specialist; (3)18 ≤ age ≤ 60 years, both gender;

(4) Patients have clear consciousness and could communicate with others normally; (5) Patients could understand the full study protocol and written informed consent is provided by themselves; (6) Those who did not use other therapies other than the basic treatment and this experimental therapy. The basic treatment refers to basic antidepressant medications under the supervision of a specialist. The basic antidepressant medications are Selective Serotonin Reuptake Inhibitors, Serotonin-Norepinephrine Reuptake Inhibitors, Norepinephrine-Dopamine Reuptake Inhibitors, Tricyclic antidepressants, Monoamine Oxidase Inhibitors. Note: Subjects who meet the above six items will be included.

Exclusion Criteria:

Exclusion criteria for healthy subjects:

1. Subjects suﬀering from mental illness, severe depression, alcohol dependence or a history of drug abuse;
2. Subjects in pregnancy, lactation or menstrual period;
3. Subjects have a fever;
4. Subjects have visible skin damage or scars in the face;
5. Subjects participating in other trials. Note: Subjects who meet any of the above will be excluded.

Exclusion criteria for MDD patients:

1. Patients with bipolar disorder;
2. Patients with schizophrenia or other mental disorders;
3. Patients with severe medical diseases, tumors or diseases of the central nervous system;
4. Patients suﬀering from severe depressive episode with psychotic symptoms;
5. Suicidal patients;
6. Patients with seasonal depression;
7. Patients with organic depression;
8. Patients with alcohol or drug addicts;
9. Patients using other therapies;
10. Patients in pregnancy or lactation;
11. Patients suffering from cognitive dysfunction, aphasia or other diseases that cannot cooperate with treatment;
12. Patients with pacemakers;
13. Patients who are not suitable for EA. Note: Subjects who meet any of the above will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Average facial temperature | Change from Baseline average facial temperature at 4 weeks
  Take the average facial temperature of 10 infrared images as the observation index, observe the change rule of the average temperature of MDD patient by comparing with healthy people.

SECONDARY OUTCOMES:
Infrared thermal images | Change from Baseline average facial temperature at 4 weeks
  Direct contrast comparisons of the approximate distribution area of the high temperature and low temperature zone of the face between healthy subjects versus MDD patients will be done using software analyses.
Hamilton depression scale (HAMD) | HAMD will be performed in the first week, the second week and the fourth week to evaluate the severity of the disease and the treatment effect.
  This scale is performed by two trained raters to perform a Hamilton depression scale (HAMD), usually in the form of conversation and observation. After the examination, the two raters will score independently. HAMD score of 21 to 35 values, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaoyu Li, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR